CLINICAL TRIAL: NCT02745041
Title: Fibrinogen Concentrate vs Cryoprecipitate in Traumatic Haemorrhage: A Pilot Randomised Controlled Trial
Brief Title: Fibrinogen Early In Severe Trauma studY
Acronym: FEISTY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gold Coast Hospital and Health Service (Other Government)
Collaborators: Emergency Medicine Foundation (Other); National Blood Authority (Other); Australian Red Cross (Other)
Responsible Party: Principal Investigator, Dr James Winearls, BSc (Hons), MBBS, MRCP, FCICM, Consultant Intensivist, GCUH ICU, Gold Coast Hospital and Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FEISTY-1
Record Dates: First submitted 2016-04-05; First posted 2016-04-20 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Trauma; Haemorrhage; Coagulopathy
Keywords: Fibrinogen; Cryoprecipitate
MeSH Terms: conditions — Wounds and Injuries; Hemorrhage; Hemostatic Disorders | interventions — Fibrinogen; cryoprecipitate coagulum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fibrinogen Concentrate (Experimental): Fibrinogen Replacement using Fibrinogen Concentrate as per ROTEM guided treatment algorithm [FIBTEM ≤ A5 10mm]
  Interventions: Drug: Fibrinogen Concentrate
- Cryoprecipitate (Active Comparator): Fibrinogen replacement using Cryoprecipitate as per ROTEM guided treatment algorithm [FIBTEM A5 ≤ 10mm]
  Interventions: Other: Cryoprecipitate

INTERVENTIONS:
Drug: Fibrinogen Concentrate — Fibrinogen Replacement using Fibrinogen Concentrate as per ROTEM guided treatment algorithm [FIBTEM ≤ A5 10mm]
  FIBTEM A5 0mm (Flat Line) = 6g FC FIBTEM A5 1 - 4mm = 5g FC FIBTEM A5 5 - 6mm = 4g FC FIBTEM A5 7 - 8mm = 3g FC FIBTEM A5 9 - 10mm = 2g FC
  Other Names: RIASTAP
  Arms: Fibrinogen Concentrate
Other: Cryoprecipitate — Fibrinogen replacement using Cryoprecipitate as per ROTEM guided treatment algorithm [FIBTEM A5 ≤ 10mm]
  FIBTEM A5 0mm (Flat Line) = 20 Units Cryo FIBTEM A5 1- 4mm = 16 Units Cryo FIBTEM A5 5 - 6mm = 14 Units Cryo FIBTEM A5 7 - 8mm = 10 Units Cryo FIBTEM A5 9 - 10mm = 8 Units Cryo
  Arms: Cryoprecipitate

SUMMARY:
* Haemorrhage in severe trauma is a significant cause of mortality and is potentially the most preventable cause of death in trauma patients
* Trauma Induced Coagulopathy (TIC) is a complex coagulopathy associated with severe trauma
* Hypo/dysfibrinogenaemia plays an important role in TIC
* Early replacement of fibrinogen may improve outcomes
* Fibrinogen replacement is potentially inadequate in standard fixed ratio Major Haemorrhage Protocols (MHP) utilising Plasma and/or Cryoprecipitate
* The majority of centres utilise cryoprecipitate for additional fibrinogen supplementation as part of a MHP
* Cryoprecipitate administration is often delayed (between 60 - 120 minutes) in a fixed ratio MHP
* It is clear early intervention in severe traumatic haemorrhage is associated with improved outcomes - CRASH 2 and PROPPR studies
* Increasing interest in the use of Fibrinogen Concentrate (FC) in severe bleeding but not supported by high level evidence
* Benefits of FC - viral inactivation, known dose, easily reconstituted, can be administered quickly in high dose and stored at room temperature in the trauma resuscitation bay
* No previous studies comparing FC and Cryoprecipitate in bleeding trauma patients
* Fibrinogen supplementation will be guided by an accepted ROTEM targeted treatment algorithm
* It will be a pilot, multi-centre randomised controlled trial comparing FC to Cryoprecipitate (current standard practise in fibrinogen supplementation)
* Hypothesis: Fibrinogen replacement in severe traumatic haemorrhage can be achieved quicker with a more predictable dose response using Fibrinogen Concentrate compared to Cryoprecipitate
* It is imperative that robust and clinically relevant trials are performed to investigate fibrinogen supplementation in trauma before widespread adoption makes performing such studies unfeasible

ELIGIBILITY:
Inclusion Criteria:

1. Adult affected by Trauma (>18yrs) and
2. Judged to have significant haemorrhage or
3. Predicted to require significant transfusion with ABC Score ≥ 2 or by treating clinician judgement

Exclusion Criteria:

1. Injury judged incompatible with survival
2. Pregnancy
3. Known objection to blood products
4. Previous Fibrinogen replacement this admission
5. Pre-Trauma Centre fibrinogen replacement
6. Participation in competing study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12; Primary Completion 2018-01-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Time to administration of Fibrinogen Replacement from time of ROTEM analysis indicating fibrinogen supplementation is required First dose of Fibrinogen Concentrate or Cryoprecipitate required | 3 Hours
  It is anticipated that fibrinogen replacement will occur with 3 hours Fibrinogen replacement will be with either FC or Cryroprecipitate depending on randomisation
Feasibility of administering FC within 30 mins of clinical scenario and ROTEM analysis suggesting Fibrinogen replacement is required | 3 Hours
  Proportion of patients receiving FC within 30 minutes
Effects on Fibrinogen levels during traumatic haemorrhage as measured by Clauss Fibrinogen | 7 Days
  Blood sampling will occur for 7 days after admission/randomisation
Effects on Fibrinogen levels during traumatic haemorrhage as measured by FIBTEM | 7 Days
  Blood sampling will occur for 7 days after admission/randomisation

SECONDARY OUTCOMES:
Transfusion Requirements | 48 hours
  In number of units of Packed Red Blood Cells, Plasma, FC, Cryoprecipitate, Platelets, Prothrombin Complex Concentrate at 4, 6, 24, 48hrs
Duration of bleeding episode or time until surgical control | 12 hours
  It is anticipated that haemorrhage control will be achieved within 12 hours
Intensive Care Unit Length of stay | 1 Year
Hospital Length of Stay | 1 Year
Adverse Events | 1Year
  Transfusion related adverse events Sepsis Multiple Organ Failure Acute Renal Failure Thromboembolic Complications
All cause Mortality | 90 Days
  Mortality at 4, 6, 24 hours and up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: James Winearls, MBBS, Principal Investigator — Gold Coast University Hospital
Locations (4):
- Australia (4):
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Townsville Hospital, Townsville, Queensland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morrow GB, Feller T, McQuilten Z, Wake E, Ariens RAS, Winearls J, Mutch NJ, Laffan MA, Curry N. Cryoprecipitate transfusion in trauma patients attenuates hyperfibrinolysis and restores normal clot structure and stability: Results from a laboratory sub-study of the FEISTY trial. Crit Care. 2022 Sep 26;26(1):290. doi: 10.1186/s13054-022-04167-x. PMID 36163263
- [Derived] Winearls J, Wullschleger M, Wake E, Hurn C, Furyk J, Ryan G, Trout M, Walsham J, Holley A, Cohen J, Shuttleworth M, Dyer W, Keijzers G, Fraser JF, Presneill J, Campbell D. Fibrinogen Early In Severe Trauma studY (FEISTY): study protocol for a randomised controlled trial. Trials. 2017 May 26;18(1):241. doi: 10.1186/s13063-017-1980-x. PMID 28549445